CLINICAL TRIAL: NCT03374618
Title: Neutrophil Extracellular Traps in Different Forms of Systemic Sclerosis
Brief Title: Neutrophil Extracellular Traps in Systemic Sclerosis
Acronym: NET-SSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO17014
Record Dates: First submitted 2017-10-06; First posted 2017-12-15 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Systemic Lupus Erythematosus; Systemic Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- systemic lupus erythematosus (Experimental): adult with systemic lupus erythematosus
  Interventions: Other: Blood sample
- systemic sclerosis (Experimental): adult with systemic sclerosis
  Interventions: Other: Blood sample
- healthy volunteers (Other): healthy volunteer (adult)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample to quantify and qualify netosis in vivo and ex vivo after different stimulations in SSC, SLA and healthy controls

SUMMARY:
Systemic sclerosis (SSC) is a systemic disease characterized by limited or diffuse cutaneous sclerosis, microangiopathy, overproduction of autoantibodies and variable organ damage due to vasculopathy and/or fibrosis. The loss of self-tolerance is believed to be caused by the dysregulation of both innate and adaptive immune systems and may involve reactive oxygen species (ROS).

Neutrophils are potent producers of ROS and may play a role in endothelial cells and fibrobasts dysfunction, as in autoantibodies generation. However, their role in SSC pathogenesis remains to be determined. Recent studies discovered abnormal regulation of neutrophil extracellular traps (NETs) in other auto-immune diseases such as systemic lupus erythematosus (SLE). NETs are web-like structures composed of chromatin backbones and granular molecules. They are released by activated neutrophils through a process called "NETosis". Nets were first described in 2004 as a novel host defense mechanism to trap and kill foreign pathogens. Recent evidence shows that NETs also participate in the pathogenesis of a variety of inflammatory and autoimmune diseases, including SLE.

We hypothesis that this phenomenon could be dysregulated in SSC as in SLE and could play a prominent role in the induction of autoimmunity, as well as in the induction and perpetuation of organ damages.

DETAILED DESCRIPTION:
This study is designed to assess the role of neutrophil extracellular traps (NETs) in systemic sclerosis as well as to evaluate the correlation between NETs production and NETs composition and the different complications and phenotypes observed in SSC.

30 SSC patients, 30 SLE patients and 60 healthy subjects will be recruited. Blood samples will be collected to obtain plasma, serum and polynuclear neutrophils by negative selection.

1. The main aim of the study is to evaluate the quantity of NETs induced by serum from SSc patients on neutrophils from either healthy or SSC patients in vitro. The quantity of NETs produced by different populations of neutrophils in contact with sera from SSC will be compared with those produced by the same different populations of neutrophils in contact with sera from SLE, and healthy subjects (two control populations).
2. Other objectives:

   * To assess the composition of the NETs produced by different populations of neutrophils exposed to serum from SSC, SLE and healthy subjects.
   * To correlate the quantity and the composition of NETS with clinical phenotype in SSc
   * To assess the role of serum cytokines in Nets production in SSC.

ELIGIBILITY:
Inclusion Criteria:

for patients of arm 1:

* patients with systemic lupus erythematosus
* patients consenting to participate to the study
* patients enrolled in the national healthcare insurance program

for patients of arm 2:

* patients with systemic sclerosis
* patients consenting to participate to the study
* patients enrolled in the national healthcare insurance program

For patients of arm 3 (healthy volunteers)

* Patients without Chronic inflammatory systemic disease
* Patients without Current or past neoplasy,
* patients without chronic metabolic pathology
* patients without treatment by anti inflammatory or corticotherapy for the last 15 days,
* patients without infectious pathology or inflammatory acute for the last 15 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Quantification of neutrophil extracellular traps (NETs) generated after stimulation of neutrophils in vitro by serum from SSC, SLE and healthy controls. | Day 0
  Comparative analysis of the quantity of neutrophil extracellular traps (NETs) generated after stimulation of neutrophils in vitro by serum from SSC, SLE and healthy controls. Neutrophils from SSC, SLE and healthy subjects will be used.

SECONDARY OUTCOMES:
Analysis of the composition of neutrophil extracellular traps | Day 0
  Comparative analysis of the composition of neutrophil extracellular traps (NETs) generated after stimulation of neutrophils in vitro by serum from SSC, SLE and healthy controls. Neutrophils from SSC, SLE and healthy subjects will be used.
Analysis of the cytokines influencing NETs production in vitro | Day 0
  Comparative analysis of the quantity of neutrophil extracellular traps (NETs) generated after stimulation of neutrophils from SSC patients in vitro by differents cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France